CLINICAL TRIAL: NCT03337022
Title: A Phase 1, Multi-center, Randomized, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CC-90006 Administered Subcutaneously in Patients With Plaque-type Psoriasis
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CC-90006 in Subjects With Mild to Moderate Plaque-type Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-90006-CP-002
Record Dates: First submitted 2017-11-07; First posted 2017-11-08 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; CC-90006; Mild to moderate plaque-type psoriasis; Safety; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CC-90006; Dose level 1 (Experimental): CC-90006 will be administered subcutaneously (SC) on days 1, 15, and 29.
  Interventions: Drug: CC-90006
- CC-90006; Dose level 2 (Experimental): CC-90006 will be administered subcutaneously (SC) on days 1, 15, and 29.
  Interventions: Drug: CC-90006
- CC-90006; Dose level 3 (Experimental): CC-90006 will be administered subcutaneously (SC) on days 1, 15, and 29.
  Interventions: Drug: CC-90006
- CC-90006; Dose level 4 (Experimental): CC-90006 will be administered subcutaneously (SC) on days 1, 15, and 29.
  Interventions: Drug: CC-90006
- Placebo (Placebo Comparator): Placebo (saline) will be administered subcutaneously (SC) on days 1, 15, and 29.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-90006 — CC-90006
  Arms: CC-90006; Dose level 1; CC-90006; Dose level 2; CC-90006; Dose level 3; CC-90006; Dose level 4
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), and immunogenicity of CC-90006 following administration of multiple subcutaneous doses in subjects with mild to moderate plaque-type psoriasis.

DETAILED DESCRIPTION:
The study will be conducted in subjects with mild to moderate plaque-type psoriasis.

The study will consist of escalating multiple (three) doses in sequential groups. Approximately 40 subjects with plaque-type psoriasis will be enrolled into approximately 4 planned dose cohorts.

Each cohort will study a different CC-90006 dose level and have ten subjects; eight subjects will receive CC-90006 and two subjects will receive placebo. Subjects will be dosed according to a computer-generated randomization scheme. Dosing will occur on Days 1, 15 (Week 2), and 29 (Week 4). During the study, blood samples and punch biopsies will be collected to determine the amount of CC-90006 in the body and to evaluate its effect on the subject's condition. Subjects will return to the clinic for regular follow up visits for safety, PK, and PD. A follow up phone call to each subject to determine general health will occur on Day 141 (week 20).

ELIGIBILITY:
Inclusion Criteria:

The following is a summary of the inclusion criteria:

1. Males or non-pregnant females between the ages of 18 and 60 years (inclusive) at the time of signing the ICF, and be willing to adhere to the requirements of contraception use throughout the study.

   1. Female subjects who claim to be surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral salpingo-oophorectomy; proper documentation required) must have undergone the procedure at least 6 months before screening,
   2. Females who claim to be postmenopausal (defined as 24 consecutive months without menses before screening, should have a confirmed follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
   3. All other females must:

   i. Have two negative pregnancy tests (at screening and baseline) as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.

   ii. Either commit to true abstinence from heterosexual contact or agree to use two forms of reliable contraception simultaneously. One must be a highly effective method and one additional effective (barrier) method, and both must be practiced without interruption, 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 4 months after discontinuation of study therapy.

   d. Males must practice true abstinence1 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP2 while participating in the study, during dose interruptions, and for at least 4 months after the last dose of IP, even if he has undergone a successful vasectomy.
2. Must be diagnosed with mild to moderate plaque-type psoriasis at least 6 months prior to baseline (Day 1).
3. Must have a PASI ≤ 15 at screening and baseline (Day 1).
4. Must have a body surface area affected score (BSA) ≥ 1 and sPGA ≥ 3 at screening and baseline (Day 1).
5. Must have at least two plaques, at least 3 x 3 centimeters(cm) in diameter. One plaque will be used for punch biopsy and the other for TPSS evaluation.
6. Other than the diagnosed condition of mild to moderate plaque-type psoriasis, the subject must be in good health as determined by a physical examination (PE) at screening.
7. Has a body mass index (BMI) ≥ 18 and ≤ 35 kg/m2 at screening.
8. For all other clinical laboratory safety test parameters, the subject has results within normal limits or judged to be not clinically significant by the Investigator.

Exclusion Criteria:

The following is a summary of the exclusion criteria:

1. Presence of any significant medical condition, laboratory abnormality, or psychiatric illness which places him or her at unacceptable risk by participating in the study, or that would that would prevent the subject from participating in the study for other reasons, or would confound the ability to interpret data from the study.
2. History of cancer.
3. Presence of cancer or pre-cancerous conditions,
4. Presence of confirmed cervical dysplasia.
5. Presence of a systemic infection or any potentially opportunistic infections (eg, atypical mycobacterial, CMV, Clostridium difficile, multifocal herpetic, etc).

   (Immunologic disorders such as rheumatoid arthritis, lupus, asthma, and any immunodeficiency are exclusionary.)
6. Presence of latent tuberculosis infection and/or active tuberculosis disease, as tested using QuantiFERON-TB Gold test (or equivalent). Subjects with a history of TB who have completed treatment (documented) may be eligible for the study.
7. History of serum hepatitis, or a confirmed carrier of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcA), or hepatitis C virus antibody (HCV Ab), or who has a positive HIV antibody test.
8. Presence of non-plaque psoriasis (erythrodermic, guttate, inverse, or pustular psoriasis).
9. Presence of dermatological diseases other than plaque psoriasis, including but not limited to seborrheic dermatitis, lichen simplex chronicus, atopic dermatitis, nummular eczema, superficial fungal infections, subacute cutaneous lupus erythematosus, pityriasis rubra pilaris, crusted scabies, cutaneous T cell lymphoma
10. Use of topical therapy for psoriasis within 14 days of first dosing (including but not limited to corticosteroids, retinoids, vitamin D analog, calcineurin inhibitors, salicylic acid).
11. Use of systemic therapy for psoriasis within 30 days of first dose administration.
12. Use of phototherapy for psoriasis within 30 days of first dose administration.
13. Use of systemic biologics treatment for psoriasis within 24 weeks of first dose administration.
14. Exposure to an immunosuppressive or immunomodulatory drug within 30 days of first dose administration, or five half-lives of the drug (whichever is longer).
15. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
16. Smoking > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
17. Vaccination within 30 days prior to the first dose administration or subject has plans to receive a vaccination during the course of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately Week 20
  Number of participants with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax | Up to approximately 16 weeks
  Observed maximum concentration of CC-90006 in serum
Pharmacokinetics - Tmax | Up to approximately 16 weeks
  Time to reach the observed maximum concentration of CC-90006 in serum
Pharmacokinetics - AUC 0-t | Up to approximately 16 weeks
  Area under that serum-concentration time curve calculated from time zero to the last measured time point
Pharmacokinetics - AUC 0-∞ | Up to approximately 16 weeks
  Area under that serum-concentration time curve calculated from time zero to ∞
Pharmacokinetics - t1/2 | Up to approximately 16 weeks
  Terminal elimination half-life
Pharmacokinetics - CL/F | Up to approximately 16 weeks
  Apparent clearance of drug from serum after extravascular administration
Pharmacokinetics - Vz/F | Up to approximately 16 weeks
  Apparent volume of distribution during the terminal phase
Pharmacokinetics - Rac [AUCτ] | Up to approximately 16 weeks
  Accumulation ratio based on Cmax (Rac [Cmax]) and AUCτ
Fraction of subjects with Anti-drug antibody (ADA) | Up to approximately 16 weeks
  Measure of the body's immune response to CC-90006

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene Corporation
Locations (4):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - TKL Research, Fair Lawn, New Jersey
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- Innovaderm Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No